CLINICAL TRIAL: NCT04961385
Title: Immunogenicity of the ChAdox1 n CoV-19 Vaccine Against SARS-CoV-2 With 12-dose Vials: an Interim Analysis
Brief Title: Immunogenicity of the ChAdox1 n CoV-19 Vaccine With 12-dose Vial
Status: Completed | Type: Observational
Sponsor: Bangkok Metropolitan Administration Medical College and Vajira Hospital (Other Government)
Responsible Party: Principal Investigator, Thananda Trakarnvanich, Associate Professor, Bangkok Metropolitan Administration Medical College and Vajira Hospital
Other Study IDs: 111/64
Record Dates: First submitted 2021-06-25; First posted 2021-07-14 (Actual); Last update posted 2021-07-14 (Actual); Status verified 2021-07

CONDITIONS: Covid19; Vaccine; Immunogenicity
Keywords: COVID-19; Immunogenicity; Neutralising antibody; Antispike RBD; ChAd0x1 nCoV-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ChAd0x1 nCoV-19 vaccinees: Participants who received first dose of ChAdox-1 n COV-19 were recruited. Participants were eligible if they were more than 18 years old
  Interventions: Biological: Immunogenicity after first dose of participants who received first dose of ChAdox-1 n COV-19 vaccine

INTERVENTIONS:
Biological: Immunogenicity after first dose of participants who received first dose of ChAdox-1 n COV-19 vaccine — Blood samples were taken from the vaccinated participants for antibody testing against SARS-CoV-2

SUMMARY:
ChAd0x1 nCoV-19 (AZD 1222) is the main vaccine that is planned to roll-out in Thailand and involve vaccinating people especially in high-risk categories. This vaccine is contained in the multiple-dose vial for vaccinating 10 recipients for 0.5 mL each. However, the additional volume of vaccine was overfilled to 6.5 mL per vial which the vaccination can be administered to more than 10 doses. The University Hospital Network (UHOSNET) and Faculty of Medicine Vajira Hospital, Navamindradhiraj University have jointly stipulated the preparation and vaccination of ChAdox1 - n CoV-19 vaccine with 12 doses per vial injection with traditional 21 or 24 G needle. Taken together, The investigators planned to investigate the immune response of participants after first dose of ChAd0x1 nCoV-19 vaccination with such technique

DETAILED DESCRIPTION:
The investigators measured anti-SARS-CoV-2 antispike RBD IgG and neutralizing antibody by surrogate virus neutralizing test (sVNT) in adults between age 18-72 year after first dose of ChAd0x1 nCoV-19 vaccine.The primary outcome was the antibody levels.The secondary outcome were adverse events,factors affecting antibody levels and incidence of COVID-19 infection at the time of study

ELIGIBILITY:
Inclusion Criteria:

* Participants were eligible if they were more than 18 years old.

Exclusion Criteria:

* Allergic to components of vaccine
* Risk of COVID-19 infection in the previous 14 days before enrollment i.e close contact with index cases or history of fever with upper respiratory tract infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants who received first dose of ChAdox-1 n COV-19 were recruited.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2021-05-31 (Actual); Study Completion 2021-05-31 (Actual)

PRIMARY OUTCOMES:
Antispike RBD IgG level | Baseline
  Level inBAU/ml
Antispike RBD IgG level | 3 monnths
  Level inBAU/ml
Antispike RBD IgG level | 6 months
  Level inBAU/ml
Neutralizing antibody | Baseline
  Percent inhibition
Neutralizing antibody | 3 months
  Percent inhibition
Neutralizing antibody | 6 months
  Percent inhibition

SECONDARY OUTCOMES:
Adverse events | through study completion,an average of 1 year
  Any abnormal symptoms post vaccination
Covid-19 infection | through study completion,an average of 1 year
  Incidence of COVID-19 infection

CONTACTS AND LOCATIONS:
Locations (1):
- Thananda Trakarnvanich, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: Yes
Mandeley website
Supporting Information: Study Protocol
Time Frame: As soon as the manuscript is accepted for publication

REFERENCES:
- [Background] Le Dare B, Bacle A, Lhermitte R, Lesourd F, Lurton Y. Maximizing number of doses drawn from multi-dose COVID-19 vaccines by minimizing dead-volume. J Travel Med. 2021 Jun 1;28(4):taab049. doi: 10.1093/jtm/taab049. No abstract available. PMID 33772277
- [Background] Kesten JM, Ayres R, Neale J, Clark J, Vickerman P, Hickman M, Redwood S. Acceptability of low dead space syringes and implications for their introduction: A qualitative study in the West of England. Int J Drug Policy. 2017 Jan;39:99-108. doi: 10.1016/j.drugpo.2016.09.005. Epub 2016 Oct 24. PMID 27788406
- [Background] Tan CW, Chia WN, Qin X, Liu P, Chen MI, Tiu C, Hu Z, Chen VC, Young BE, Sia WR, Tan YJ, Foo R, Yi Y, Lye DC, Anderson DE, Wang LF. A SARS-CoV-2 surrogate virus neutralization test based on antibody-mediated blockage of ACE2-spike protein-protein interaction. Nat Biotechnol. 2020 Sep;38(9):1073-1078. doi: 10.1038/s41587-020-0631-z. Epub 2020 Jul 23. PMID 32704169
- [Result] Strauss K, van Zundert A, Frid A, Costigliola V. Pandemic influenza preparedness: the critical role of the syringe. Vaccine. 2006 May 29;24(22):4874-82. doi: 10.1016/j.vaccine.2006.02.056. Epub 2006 Mar 20. PMID 16647790
- [Result] Mehran R, Dangas GD, Weisbord SD. Contrast-Associated Acute Kidney Injury. N Engl J Med. 2019 May 30;380(22):2146-2155. doi: 10.1056/NEJMra1805256. No abstract available. PMID 31141635
- [Result] Folegatti PM, Ewer KJ, Aley PK, Angus B, Becker S, Belij-Rammerstorfer S, Bellamy D, Bibi S, Bittaye M, Clutterbuck EA, Dold C, Faust SN, Finn A, Flaxman AL, Hallis B, Heath P, Jenkin D, Lazarus R, Makinson R, Minassian AM, Pollock KM, Ramasamy M, Robinson H, Snape M, Tarrant R, Voysey M, Green C, Douglas AD, Hill AVS, Lambe T, Gilbert SC, Pollard AJ; Oxford COVID Vaccine Trial Group. Safety and immunogenicity of the ChAdOx1 nCoV-19 vaccine against SARS-CoV-2: a preliminary report of a phase 1/2, single-blind, randomised controlled trial. Lancet. 2020 Aug 15;396(10249):467-478. doi: 10.1016/S0140-6736(20)31604-4. Epub 2020 Jul 20. PMID 32702298
- [Result] Voysey M, Clemens SAC, Madhi SA, Weckx LY, Folegatti PM, Aley PK, Angus B, Baillie VL, Barnabas SL, Bhorat QE, Bibi S, Briner C, Cicconi P, Collins AM, Colin-Jones R, Cutland CL, Darton TC, Dheda K, Duncan CJA, Emary KRW, Ewer KJ, Fairlie L, Faust SN, Feng S, Ferreira DM, Finn A, Goodman AL, Green CM, Green CA, Heath PT, Hill C, Hill H, Hirsch I, Hodgson SHC, Izu A, Jackson S, Jenkin D, Joe CCD, Kerridge S, Koen A, Kwatra G, Lazarus R, Lawrie AM, Lelliott A, Libri V, Lillie PJ, Mallory R, Mendes AVA, Milan EP, Minassian AM, McGregor A, Morrison H, Mujadidi YF, Nana A, O'Reilly PJ, Padayachee SD, Pittella A, Plested E, Pollock KM, Ramasamy MN, Rhead S, Schwarzbold AV, Singh N, Smith A, Song R, Snape MD, Sprinz E, Sutherland RK, Tarrant R, Thomson EC, Torok ME, Toshner M, Turner DPJ, Vekemans J, Villafana TL, Watson MEE, Williams CJ, Douglas AD, Hill AVS, Lambe T, Gilbert SC, Pollard AJ; Oxford COVID Vaccine Trial Group. Safety and efficacy of the ChAdOx1 nCoV-19 vaccine (AZD1222) against SARS-CoV-2: an interim analysis of four randomised controlled trials in Brazil, South Africa, and the UK. Lancet. 2021 Jan 9;397(10269):99-111. doi: 10.1016/S0140-6736(20)32661-1. Epub 2020 Dec 8. PMID 33306989
- [Result] Ramasamy MN, Minassian AM, Ewer KJ, Flaxman AL, Folegatti PM, Owens DR, Voysey M, Aley PK, Angus B, Babbage G, Belij-Rammerstorfer S, Berry L, Bibi S, Bittaye M, Cathie K, Chappell H, Charlton S, Cicconi P, Clutterbuck EA, Colin-Jones R, Dold C, Emary KRW, Fedosyuk S, Fuskova M, Gbesemete D, Green C, Hallis B, Hou MM, Jenkin D, Joe CCD, Kelly EJ, Kerridge S, Lawrie AM, Lelliott A, Lwin MN, Makinson R, Marchevsky NG, Mujadidi Y, Munro APS, Pacurar M, Plested E, Rand J, Rawlinson T, Rhead S, Robinson H, Ritchie AJ, Ross-Russell AL, Saich S, Singh N, Smith CC, Snape MD, Song R, Tarrant R, Themistocleous Y, Thomas KM, Villafana TL, Warren SC, Watson MEE, Douglas AD, Hill AVS, Lambe T, Gilbert SC, Faust SN, Pollard AJ; Oxford COVID Vaccine Trial Group. Safety and immunogenicity of ChAdOx1 nCoV-19 vaccine administered in a prime-boost regimen in young and old adults (COV002): a single-blind, randomised, controlled, phase 2/3 trial. Lancet. 2021 Dec 19;396(10267):1979-1993. doi: 10.1016/S0140-6736(20)32466-1. Epub 2020 Nov 19. PMID 33220855